CLINICAL TRIAL: NCT02824263
Title: Metabolic Impact of Intermittent CPAP
Acronym: MIIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Academy of Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00086830; R01HL135483 (NIH)
Record Dates: First submitted 2016-03-18; First posted 2016-07-06 (Estimated); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; CPAP; metabolism
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Usual care) (No Intervention): Continuation of established CPAP therapy. CPAP will be worn during a metabolic sleep study in the research laboratory.
- CPAP withdrawal; (Experimental): Cessation of established CPAP therapy for 3 nights. CPAP will NOT be worn during this period, and a metabolic sleep study off CPAP is performed in the research laboratory on the third night.
  Interventions: Other: CPAP withdrawal

INTERVENTIONS:
Other: CPAP withdrawal — CPAP is discontinued for 3 nights.
  Arms: CPAP withdrawal;

SUMMARY:
Obstructive sleep apnea is a risk factor for diabetes and cardiovascular disease, by unknown mechanisms. The investigators hypothesize that sleep apnea changes glucose and lipid metabolism during sleep, which over time could lead to diabetes and cardiovascular disease. This study examines metabolic changes during sleep in patients with obstructive sleep apnea. Patients accustomed to continuous positive airway pressure (CPAP) therapy are enrolled to undergo sleep studies, either on CPAP therapy or after withdrawing from CPAP for 3 nights. During sleep, blood samples are obtained so that metabolic function can be compared between sleep apnea and CPAP nights.

DETAILED DESCRIPTION:
Participants with a history of moderate severe sleep apnea (AHI>20) will be enrolled if participants meet inclusion/exclusion criteria. Investigators will report to the sleep laboratory on two nights, (1) after continuing their CPAP or (2) after discontinuing CPAP for 3 nights. The order of observation will be randomized. A standard research dinner is provided before each study. IV's are placed so that blood can be sampled at frequent (30 min) intervals throughout the night. In the morning after each study, a glucose tolerance test and endothelial function study (endoPAT) are performed. Serum samples will be analyzed for glucose, insulin, free fatty acids, triglycerides, hormones, and other metabolic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* History of moderate to severe Obstructive sleep apnea (OSA) (AHI or respiratory disturbance index (RDI)> 10).
* They must also own a CPAP machine and report the ability to tolerate sleeping with or without CPAP during the night.

Exclusion Criteria:

* Uncontrolled hypertension with systolic blood pressure >170 or diastolic blood pressure > 110
* Congestive heart failure
* Use of clonidine or nicotinic acid medication
* Diabetes requiring the use of insulin
* Known pregnancy, by urine testing in women of child-bearing age
* History of falling asleep while driving, near miss
* High risk occupation (pilot, commercial driver)
* Hemoglobin < 10 g/dL on point of care screening

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chopra S, Rathore A, Younas H, Pham LV, Gu C, Beselman A, Kim IY, Wolfe RR, Perin J, Polotsky VY, Jun JC. Obstructive Sleep Apnea Dynamically Increases Nocturnal Plasma Free Fatty Acids, Glucose, and Cortisol During Sleep. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3172-3181. doi: 10.1210/jc.2017-00619. PMID 28595341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a history of obstructive sleep apnea (OSA) who were accustomed to CPAP use were enrolled from the Johns Hopkins Sleep Disorders Center.
Pre-assignment Details: 144 participants signed a consent form. 15 subjects withdrew or were lost to follow up after consent, leaving 129 participants who were randomized to CPAP first (61) or CPAP withdrawal first (68) visits.
Groups:
- CPAP First, Then OSA (CPAP Withdrawal): This is a crossover study comparing effects of sleep apnea (CPAP withdrawal) vs CPAP.
  Participants first underwent a CPAP study (continuation of established CPAP therapy) during 1 overnight visit in the sleep lab. After a washout of 1 to 4 weeks, they then had a OSA (CPAP withdrawal) study during 1 overnight visit in the sleep lab.
- OSA First (CPAP Withdrawal), Then CPAP: This is a crossover study comparing effects of sleep apnea (CPAP withdrawal) vs CPAP.
  Participants first underwent an OSA (CPAP withdrawal) study during 1 overnight visit in the sleep lab. After a washout of 1 to 4 weeks, they then had a CPAP (continuation of established CPAP therapy) study during 1 overnight visit in the sleep lab.
Period: First Intervention (1 Night)
Arm/Group | CPAP First, Then OSA (CPAP Withdrawal) | OSA First (CPAP Withdrawal), Then CPAP
Started | 61 | 68
Completed | 61 | 68
Not Completed | 0 | 0
Period: Washout (1 to 4 Weeks)
Arm/Group | CPAP First, Then OSA (CPAP Withdrawal) | OSA First (CPAP Withdrawal), Then CPAP
Started | 61 | 68
Completed | 59 | 62
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 2 | 6
Period: Second Intervention (1 Night)
Arm/Group | CPAP First, Then OSA (CPAP Withdrawal) | OSA First (CPAP Withdrawal), Then CPAP
Started | 59 | 62
Completed | 55 | 59
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: 144 participants signed a consent form, but 15 were lost to follow up before visit 1. Therefore the baseline characteristics reflect 129 participants who had demographic information collected.
Groups:
- CPAP First, Then OSA (CPAP Withdrawal): This is a crossover study comparing effects of sleep apnea (CPAP withdrawal) vs CPAP.
  Participants in this arm undergo a (1) CPAP study (continuation of established CPAP therapy), followed by a (2) CPAP withdrawal study.
- OSA First (CPAP Withdrawal), Then CPAP: This is a crossover study comparing effects of sleep apnea (CPAP withdrawal) vs CPAP.
  Participants in this arm undergo a (1) CPAP withdrawal study, followed by a (2) CPAP study (continuation of established CPAP therapy).
- Total: Total of all reporting groups
Arm/Group | CPAP First, Then OSA (CPAP Withdrawal) | OSA First (CPAP Withdrawal), Then CPAP | Total
Number analyzed (Participants) | 61 | 68 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 53 (12) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 40 | 42 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 60 | 65 | 125
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 21 | 17 | 38
  Race: Asian | 4 | 2 | 6
  Race: Caucasian | 35 | 44 | 79
  Race: Mixed | 1 | 4 | 5
  Race: Native American | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 68 | 129
Diabetes status [Count of Participants; unit: Participants]
  No diabetes | 25 | 34 | 59
  Prediabetes | 17 | 11 | 28
  Diabetes | 19 | 23 | 42
History of hypertension [Count of Participants; unit: Participants]
  Hypertension | 31 | 31 | 62
  No hypertension | 30 | 37 | 67

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Plasma Free Fatty Acids (FFA, mmol/L)
Description: We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart. Data from each night was averaged to report a single value.
Population: missing values due to IV issues leading to incomplete collection.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- CPAP; CPAP Withdrawal: This is a crossover study comparing effects of sleep apnea (CPAP withdrawal) vs CPAP.
  Participants are randomized to two arms. Either CPAP (continuation of established CPAP therapy), followed by a CPAP withdrawal
  OR
  CPAP withdrawal, followed by CPAP (continuation of established CPAP therapy)
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 109 | 109
mmol/L | 0.47 (14) | 0.51 (0.12)

2. Primary Outcome: Concentration of Plasma Glucose (mg/dl)
Description: We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart. Data from each night was averaged to report a single value.
Population: missing values due to IV issues leading to incomplete collection.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 109 | 109
mg/dl | 100 (18) | 101 (21)

3. Primary Outcome: Concentration of Plasma Insulin (mcU/ml)
Description: We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart. Data from each night was averaged to report a single value.
Population: missing values due to IV issues leading to incomplete collection.
Measure: Mean (Standard Deviation); unit: microunits/mL
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 110 | 110
microunits/mL | 18 (8) | 18 (12)

4. Primary Outcome: Concentration of Plasma Triglycerides (mg/dl)
Description: We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart. Data from each night was averaged to report a single value.
Population: Missing values due to IV issues leading to incomplete collection.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 108 | 108
mg/dl | 127 (65) | 128 (74)

5. Secondary Outcome: Oral Glucose Tolerance Test (OGTT)
Description: We will report the mean of the area under the curve (AUC) during OGTT for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart. 5 OGTT values were averaged to a obtain a single value.
Population: Missing values due to IV issues leading to incomplete collection.
Measure: Mean (Standard Deviation); unit: mg/dl*min
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 105 | 105
mg/dl*min | 19820 (5818) | 19224 (5324)

6. Secondary Outcome: Reactive Hyperemia Index (RHI)
Description: Measured in the morning using Itamar EndoPAT device. This will measure the ratio of blood flow after brachial artery occlusion to blood flow prior to brachial artery occlusion. Normal values range from approximately 1 to 3 with higher values being associated with better vascular function. We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart, 1 measurement each visit
Population: Some missing data due to technical problems during collection of EndoPAT data.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 111 | 111
Ratio | 2.21 (0.57) | 2.12 (0.65)

7. Secondary Outcome: Augmentation Index (AI)
Description: Measured in the morning using Itamar EndoPAT device. Augmentation index is measured once during each visit, and is expressed as a % increase in the pressure waveform during systole. We will report the mean for all participants per group (CPAP vs. CPAP withdrawal).
Time Frame: 2 nights, <1 month apart, 1 measurement each visit
Population: Some missing data due to technical problems during collection of EndoPAT data.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CPAP | CPAP Withdrawal
Number analyzed (Participants) | 108 | 108
percentage | 3.3 (16) | 6.3 (16)

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events beginning 3 days before each visit to screen for drowsiness related incidents. The longest duration for assessing adverse events was approximately 4 weeks (if visits 1 and 2 were 1 month apart).
Description: The risks of the study are related to IV access, temporary discontinuation of CPAP for 3 nights resulting in possible drowsiness-related incidents
Arm/Group | CPAP | CPAP Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/129
Other Adverse Events (participants affected / at risk) | 2/129 | 0/129
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (N=129) | CPAP Withdrawal (N=129)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood pressure elevation (Cardiac disorders) | 1 (1) | 0 (0) — was related to non-study related changes to medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02824263/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT02824263/ICF_001.pdf